CLINICAL TRIAL: NCT04578574
Title: Effects of Bodily Illusion and tDCS on Spinal Cord Injury (SCI) Related Neuropathic Pain
Brief Title: Effects of Bodily Illusion and tDCS on SCI-related Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida (Other)
Responsible Party: Principal Investigator, Eva Widerstrom-Noga, Research Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20200841
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BI-TDCS Stimulation Group (Experimental): Participants in this group will receive the BI and TDCS interventions for 10 sessions over two weeks.
  Interventions: Other: Bodily Illusions (BI) Procedure; Device: Transcranial direct electrical stimulation (tDCS)
- BI-TDCS (Sham) Stimulation Group (Sham Comparator): Participants in this group will receive the BI and TDCS (Sham) interventions for 10 sessions over two weeks.
  Interventions: Other: Bodily Illusions (BI) Procedure; Other: Sham Transcranial Direct Electrical Stimulation (tDCS)

INTERVENTIONS:
Other: Bodily Illusions (BI) Procedure — Each sessions will consists of two types of illusions that are 15 min each, the rubber hand illusion (RHI) and the walking illusion (WI) that involve both arms and legs.
Device: Transcranial direct electrical stimulation (tDCS) — Each sessions will consists of electrical current delivered from a battery-driven, constant current stimulator using saline-soaked surface sponge electrodes. One electrode will be placed on your scalp on the right side and the other electrode over the left eye on your forehead. A weak current will be applied for 30 min at the same time as the BI.
  Arms: BI-TDCS Stimulation Group
Other: Sham Transcranial Direct Electrical Stimulation (tDCS) — Each session of the Sham tDCS will be applied for 30 min at the same time as the BI.
  Arms: BI-TDCS (Sham) Stimulation Group

SUMMARY:
The purpose of this study is to evaluate the effect of a combination of two procedures: (1) Bodily Illusion (BI) and (2) Transcranial direct electrical stimulation (tDCS) on neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be men or women, 18-70 years of age, with an incomplete cervical traumatic SCI.
2. Participants must have experienced neuropathic pain for a minimum of six months. They must have neuropathic pain in the moderate to severe category, which will be defined as a score of at least 4 on a Numeric Rating Scale (NRS); (range of 0 to 10).
3. Participants must be willing and able to sign informed consent

Exclusion Criteria:

1. Major psychiatric disease/disorder (self-reported)
2. A significant neurological trauma besides SCI
3. A recent (one-year) history of alcohol or drug abuse (selfreported)
4. Any other medical conditions in which transcranial DCS is relatively contraindicated, such as pregnancy, epilepsy and/or seizures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Widerstrom-Noga, Phd, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BI Transcranial Direct Current Stimulation (TDCS) Stimulation Group: Participants in this group will receive the BI and TDCS interventions for 10 sessions over two weeks.
  Bodily Illusions (BI) Procedure: Each sessions will consists of two types of illusions that are 15 min each, the rubber hand illusion (RHI) and the walking illusion (WI) that involve both arms and legs.
  Transcranial direct electrical stimulation (tDCS): Each sessions will consists of electrical current delivered from a battery-driven, constant current stimulator using saline-soaked surface sponge electrodes. One electrode will be placed on your scalp on the right side and the other electrode over the left eye on your forehead. A weak current will be applied for 30 min at the same time as the BI.
Period: Overall Study
Arm/Group | BI Transcranial Direct Current Stimulation (TDCS) Stimulation Group | BI-TDCS (Sham) Stimulation Group
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BI-TDCS Stimulation Group | BI-TDCS (Sham) Stimulation Group | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (16) | 40 (7) | 48 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  White | 3 | 0 | 3
  Black American | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7
  South America | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropathic Pain Severity
Description: Assessed by the use of the Neuropathic Pain Symptom Inventory (NPSI). The NPSI has a total score ranging from 0 to 100 with the higher score indicating greater pain.
Time Frame: baseline, up to two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BI-TDCS Stimulation Group | BI-TDCS (Sham) Stimulation Group
Number analyzed (Participants) | 6 | 2
score on a scale | -7.3 (3.9) | 8.5 (6.3)

2. Primary Outcome: Change in Performance of Body Part Processing
Description: Assessed by a customized computer task, where individual reaction times will be measured in response to mental rotation of body parts. Results will be reported in milliseconds.
Time Frame: baseline, up to two weeks
Measure: Mean (Standard Deviation); unit: milliseconds (reaction times)
Arm/Group | BI-TDCS Stimulation Group | BI-TDCS (Sham) Stimulation Group
Number analyzed (Participants) | 6 | 2
milliseconds (reaction times)
  change scores in mental rotation of body parts | -18.2 (67.5) | 30.9 (25)
  change scores in mental rotation of control stimuli | -4.5 (92) | 4.4 (54)

3. Secondary Outcome: Change in Sensory Thresholds
Description: Assessed by the Quantitative Sensory Testing. Pain thresholds are evaluated using Medoc machine (Medoc Ltd,Ramat Yishai, Israel and FDA approved. It assesses participants' ability to feel change in temperature (0°C to 50°C). The temperatures in this range may be felt as cool, cold, warm, and hot. A probe is placed on the skin and it feels either cool, cold, warm or hot. Participants' thresholds are recorded for cool or warm sensation, and for cold or hot painful thresholds.
Time Frame: baseline, up to two weeks
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | BI-TDCS Stimulation Group | BI-TDCS (Sham) Stimulation Group
Number analyzed (Participants) | 6 | 2
Celsius
  delta pain threshold and perception threshold of painful site expressed as change score (hot-warm) | 2.2 (6.5) | -1.3 (4)
  delta pain thresh. and perception threshold of painful site expressed as change score (cold-cool) | -1.37 (5.4) | 3.9 (1)

ADVERSE EVENTS:
Time Frame: 1 year (during data collection)
Arm/Group | BI-TDCS Stimulation Group | BI-TDCS (Sham) Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT04578574/Prot_SAP_001.pdf